CLINICAL TRIAL: NCT03707574
Title: NCORP Tissue Procurement Protocol: An NCI Cancer Moonshot Study
Brief Title: Genetic Analysis of Blood and Tissue Samples From Patients With Advanced Cancer, Moonshot Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCI-2018-01375; NCI-2018-01375 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10231 (Other: National Cancer Institute); 10231 (Other: CTEP)
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Neoplasm; Advanced Melanoma; Advanced Renal Cell Carcinoma; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIA Ovarian Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIA1 Ovarian Cancer AJCC v8; Stage IIIA2 Ovarian Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIB Ovarian Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IIIC Ovarian Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8; Stage IVB Ovarian Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-correlative (genetic analysis): Patients undergo collection of blood and tumor prior to starting treatment and upon disease progression (second collection of blood and tumor only for patients who do not continue to progress and achieve either an OR or SD after 6 months of treatment). Samples are banked and analyzed via next generation sequencing.
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and tissue
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This trial studies the genetic analysis of blood and tissue samples from patients with cancer that has spread to other anatomic sites (advanced) or is no longer responding to treatment. Studying these samples in the laboratory may help doctors to learn how genes affect cancer and how they affect a person's response to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To procure paired newly acquired tumor tissues and blood at baseline and upon progression in patients treated for advanced cancer with molecularly targeted therapies at National Cancer Institute Community Oncology Research Program (NCORP) sites.

II. To bank formalin-fixed, paraffin-embedded (FFPE) tissue, blood (for cell-free deoxyribonucleic acid [DNA] analysis), and nucleic acids from patients in the Biorepository, which is the Biopathology Center (BPC) at Nationwide Children's Hospital (NCH), that may be used to study mechanisms of sensitivity and resistance to cancer therapies.

III. To bank, when available, optional snap-frozen tissue (for future to be determined analysis) from patients in the Biorepository, which is the Biopathology Center (BPC) at Nationwide Children's Hospital (NCH), that may be used to study mechanisms of sensitivity and resistance to cancer therapies.

IV. To assess the feasibility of obtaining paired high-quality newly acquired tumor tissues and blood from patients being treated for advanced cancer in community-based healthcare settings (NCORP sites).

SECONDARY OBJECTIVES:

I. To perform molecular profiling assays on matched malignant tumor and blood (including but not limited to whole exome and messenger ribonucleic acid [RNA] sequencing) in order to provide physicians and patients with a clinical report from a Clinical Laboratory Improvement Act (CLIA)-certified laboratory from tumor obtained at baseline and upon progression that may be used to guide further treatment planning.

II. To make available biospecimens for studies to define potential resistance biomarkers using genomic and proteomic-based assessment platforms.

III. To contribute genetic analysis data from coded specimens to Genomic Data Commons, a well annotated cancer molecular and clinical data repository, for current and future research; specimens will be annotated with key clinical data including presentation, diagnosis, staging, summary treatment, and outcome, if possible.

IV. To identify potential predictive and prognostic biomarkers beyond any genomic alteration by which treatment may be assigned.

V. To identify resistance mechanisms using genomic DNA- and RNA-based assessment platforms.

OUTLINE:

Patients undergo collection of blood and tumor prior to starting treatment and upon disease progression (second collection of blood and tumor only for patients who do not continue to progress and achieve either an objective response [OR] or stable disease [SD] after 6 months of treatment). Samples are banked and analyzed via next generation sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets all eligibility criteria for treatment of the tumors with the agents listed and has agreed to provide tissue and blood samples for this study

  * Targeted therapy maybe as a singular/monotherapy or in combination with any Food and Drug Administration (FDA)-approved chemotherapies
  * Patient's primary or recurrent disease is targeted-treatment naive or will be treated with a targeted therapy listed different from any previously-received targeted therapy or combination therapy as standard of care
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1. Patients with a PS of 2 may be enrolled only at the discretion of the treating physician and radiologist
* Have an advanced malignancy being treated with one of the agents listed. Advanced cancer is cancer that is unlikely to be cured or controlled with treatment. The cancer may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body. Treatment may be given to help shrink the tumor, slow the growth of cancer cells, or relieve symptoms. Patients may be undergoing first or subsequent lines of therapy. In the case where an agent not listed is newly approved for one of the listed tumors, patients undergoing therapy with it will be able to enroll at discretion of the principal investigator (PI). This is to avoid any lag between FDA approval of a previously investigational agent and protocol modifications/updates
* Have an advanced malignancy that meets one of the following criteria:

  * Patients must have tumor amenable to image guided or direct vision biopsy and be willing and able to undergo a tumor biopsy for molecular profiling. The biopsy must not be associated with a significant risk of severe or major complications or death. In particular, endoscopic, open or laparoscopic surgical procedures are not to be performed to provide research specimens. However, research specimens may be provided if the patient needs to undergo such procedures for clinical reasons
  * Severe or major complications are considered to be those

    * Requiring therapy, minor hospitalization (more than overnight but < 48 hours [h])
    * Requiring major therapy; unplanned increase in level of care, prolonged hospitalization > 48 h
    * Resulting in permanent adverse sequelae
    * Resulting in death
  * Patient will be undergoing a procedure due to medical necessity during which the tissue may be collected. The following tumors may be collected only under the conditions specified and not for the sole purpose of the clinical trial:

    * Brain biopsies: ONLY if the patient has medical necessity for craniotomy for clinical care
    * Mediastinal, laparoscopic, gastrointestinal, or bronchial endoscopic biopsies: ONLY to be obtained incidentally to a clinically necessary procedure

Exclusion Criteria:

* Uncontrolled intercurrent illness that in the physician's assessment would pose undue risk for biopsy
* Patients currently enrolled or planning to be co-enrolled (while participating on the 10231 study) on a therapeutically interventional clinical trial aimed to treat the current malignancy
* If the patient is on chronic anticoagulation treatment, they must be able and willing to have this treatment discontinued for the biopsy. Discontinuation procedures will be those of the treating site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for advanced cancer with molecularly targeted therapies at NCORP sites
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2026-01-23 (Actual)

PRIMARY OUTCOMES:
Obtaining tumor tissue and blood specimens | Up to 2 years
  Will obtain tumor tissue and blood specimens for biobanking and to store tissues, blood, and nucleic acids for future research, including the study of matched pre and post-treatment tumor biopsies to elucidate mechanisms of resistance. Cases will be grouped according to histology and/or treatment.

SECONDARY OUTCOMES:
Tumor tissues storage in the Biopathology Center (BPC) at Nationwide Children's Hospital (NCH) (Biorepository) | Up to 2 years
Genomic analysis | Up to 2 years
  Will perform genomic studies, including a pan-cancer gene panel, and contribute molecular data to the genomic data commons.

CONTACTS AND LOCATIONS:
Overall Officials: S. P Ivy, Principal Investigator — National Cancer Institute (NCI)
Locations (144):
- United States (143):
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - East Jefferson General Hospital, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Mercy Medical Center, Springfield, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- Doctors Cancer Center, Manatí, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm